CLINICAL TRIAL: NCT03006900
Title: Determining the Impact of a Pilates Program in Multiple Sclerosis
Brief Title: Multiple Sclerosis and Pilates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Multiple Sclerosis Society of Canada (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2918
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise Movement Techniques; Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pilates and massage (Experimental): Pilates (twice per week for 50 minutes) and massage (once per week for one hour)
  Interventions: Other: Pilates; Other: Massage
- Massage (Active Comparator): Massage (once per week for one hour)
  Interventions: Other: Massage

INTERVENTIONS:
Other: Pilates — Pilates
  Arms: Pilates and massage
Other: Massage — Massage

SUMMARY:
Pilates is becoming popular among the multiple sclerosis (MS) community as an alternative to the more traditional exercise programs. Although somewhat limited, previous research has suggested Pilates may have some beneficial effects in MS. This 12-week, single-blinded, randomized controlled study has one intervention group (Pilates and massage therapy) and one control group (massage therapy only). The primary outcome of interest is the change in walking ability between groups. Secondary outcomes include other measures of physical performance and quality of life.

DETAILED DESCRIPTION:
In the recent 2015 MS Society of Canada MS Wellness Survey almost 25% of people indicated that they think physical activity is the most important area of wellness, yet physical inactivity is still common in individuals with multiple sclerosis (MS). While some of this may be due to factors related to MS such as fatigue, pain, and physical restrictions, research has shown that exercise has beneficial effects on mobility, strength, balance, and overall quality of life. However, because the symptoms of MS vary, there is not one optimal exercise program that exists. Pilates may be a good exercise option for MS. Pilates focuses on body positions and movement, with specific attention on the core (stomach or trunk) muscles. Very few researchers have studied Pilates in MS, but those that have, noticed some improvements in walking, balance, and strength. There were no negative effects reported from the Pilates exercises, and the exercises can be adapted for all levels of ability in MS. We are interested in studying the effect of Pilates in MS. To do this, we will recruit 30 people with MS to participate in this study. Participants will be randomly put into either the Pilates group or the control group. Those individuals in the Pilates group will attend two 50-minute Pilates classes twice weekly, plus receive a weekly 1-hour massage therapy session. Individuals in the control group will only receive the weekly massage therapy session. At the end of the study (12 weeks), we will look to see if there are any differences between the two groups in walking ability. We will also compare other important outcomes such as muscle strength, balance, and quality of life between the two groups. Results from this study may provide individuals with another exercise option to help manage their MS and improve their wellness. Results will also be useful for organizations such as the MS Society to help make decisions about which programs and services to offer to individuals with MS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis

Exclusion Criteria:

* Expanded Disability Status Scale of 8 or higher

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in distance during the 6-minute walk test | 12 weeks

SECONDARY OUTCOMES:
Change from baseline in balance score for the Fullerton Advanced Balance Scale | 12 weeks
Change in sit and reach test score for flexibility | 12 weeks
Change from baseline in timed up and go test score | 12 weeks
Change from baseline in physical activity level | 12 weeks
Change from baseline in maximal isometric knee extension strength | 12 weeks
Change from baseline in ability to recruit motor units | 12 weeks
Change from baseline in ability to recruit motor units in a fatigued state | 12 weeks
Change from baseline in trunk muscular endurance | 12 weeks
Change from baseline in lean tissue mass | 12 weeks
Change from baseline in fat mass | 12 weeks
Change from baseline for score from the MS International Quality of Life questionnaire | 12 weeks
Change from baseline in adverse events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Charity Evans, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- College of Kinesiology, University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No